CLINICAL TRIAL: NCT06524362
Title: Effect of Pelvic Rehabilitation After Low Anterior Resection for Cancer Rectum. - A Randomised Controlled Trial (PERECARE TRIAL)
Brief Title: Effect of Pelvic Rehabilitation After Low Anterior Resection for Cancer Rectum. - A Randomised Controlled Trial
Acronym: PERECARE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GEM Hospital & Research Center (Other)
Collaborators: JOGO Health Pvt Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: PERECARE
Record Dates: First submitted 2024-07-23; First posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Rectal Cancer; Rectum Neoplasm; Rectal Neoplasms; Rectal Adenocarcinoma; Low Anterior Resection Syndrome; Fecal Incontinence; Bowel Dysfunction
Keywords: Pelvic Floor Rehabilitation; Low Anterior Resection; Ultra Low Anterior Resection; Rectal Cancer Surgery; Post operative care; Bowel function; Quality of life; Randomized controlled trial; Fecal Urgency; Pelvic Floor Muscle Training; Oncological outcomes
MeSH Terms: conditions — Rectal Neoplasms; Low Anterior Resection Syndrome; Fecal Incontinence; Intestinal Diseases

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pelvic Floor Physiotherapy (PFR) group (Experimental): Patients completing three months post-low anterior resection (LAR) for rectal cancer or six weeks post-diversion ileostomy closure following LAR will be recruited to Pelvic Floor Rehabilitation (PFR) group after randomization.
  Intervention: Participants will undergo a structured pelvic floor physiotherapy program for three months.
  The program includes:
  Eight Personal Sessions: Each session lasts 45 minutes.
  Frequency:
  * Once a week for the first month (four sessions).
  * Biweekly for the next two months (four sessions).
  Home Exercises: Participants will be guided on pelvic floor exercises to be performed at home throughout the three months.
  Usual Care: In addition to the pelvic floor rehabilitation, participants will receive the standard postoperative care for rectal cancer surgery.
  Interventions: Behavioral: Pelvic Floor Physiotherapy (PFR)
- Conventional group (Active Comparator): Patients completing three months post-low anterior resection (LAR) for rectal cancer or six weeks post-diversion ileostomy closure following LAR will be recruited to Conventional group after randomization.
  Recruited subjects in the conventional group recieves usual care following low anterior resection such as fluid intake, fiber intake, diet, toilet posture, life style advice etc
  Interventions: Behavioral: Conventional group

INTERVENTIONS:
Behavioral: Pelvic Floor Physiotherapy (PFR) — Intervention: Participants will undergo a structured pelvic floor physiotherapy program for three months.
  The program includes:
  Eight Personal Sessions: Each session lasts 45 minutes.
  Frequency:
  Once a week for the first month (four sessions). Biweekly for the next two months (four sessions). Home Exercises: Participants will be guided on pelvic floor exercises to be performed at home throughout the three months.
  Arms: Pelvic Floor Physiotherapy (PFR) group
Behavioral: Conventional group — Patients completing three months post-low anterior resection (LAR) for rectal cancer or six weeks post-diversion ileostomy closure following LAR will be recruited to Conventional group after randomization.
  Recruited subjects in the conventional group recieves usual care following low anterior resection such as fluid intake, fiber intake, diet, toilet posture, life style advice etc
  Arms: Conventional group

SUMMARY:
Study Purpose:

This study aims to understand how pelvic floor rehabilitation (PFR) after low anterior resection (LAR) surgery for rectal cancer affects bowel control and quality of life compared to usual care.

Background:

Rectal cancer and its treatments can significantly impact patients' lives, often causing bowel issues like frequent bowel movements, urgency, and incontinence. These problems, known as low anterior resection syndrome (LARS), affect 70-90% of patients and can last for over two years. (1,2)

Current Knowledge:

Advances in treatments have improved survival rates and recovery. Despite improvements, many patients still experience bowel issues after surgery.

Past studies show PFR can help, but they have limitations like small sample sizes and varied methods. (3-5)

Need for the Study:

There is a need for a well-designed study to confirm the benefits of PFR and to identify which patients benefit the most.

Study Design:

This study is a randomized controlled trial that will:

* Compare PFR to usual care in patients after LAR surgery.
* Focus on bowel control and quality of life.
* Provide detailed insights to improve aftercare for rectal cancer patients.

DETAILED DESCRIPTION:
This study will investigate the effects of pelvic floor rehabilitation (PFR) on bowel function and quality of life in patients who have undergone low anterior resection (LAR) for rectal cancer. The study aims to provide a more comprehensive understanding of effective aftercare for these patients. Here are the key components of the study protocol:

Study Design

Type: Randomized controlled trial.

Participants: Patients who have undergone LAR for rectal cancer.

Interventions: Pelvic floor rehabilitation compared to usual care.

Primary Outcomes: Fecal incontinence.

Secondary Outcomes: Quality of life, LARS score.

Procedures. Screening and Enrollment: Pateint with rectal cancer undergoing sphincter preserving surgeries and who are willing to participate will be enrolled after thorugh explaination of the study.

Randomization: Post three months following Low anterior resection or post 6 weeks following closure of diversion ileostomy, participants will be randomly assigned to either the PFR group or the usual care group using computer generated randomization.

Intervention: The PFR group will receive a structured pelvic floor rehabilitation program by a trained pelvic physiotherapist along with usual care. The PFR program includes three components:

1. Pelvic Floor Muscle Training: Focused on increasing maximum strength, extending contraction duration, and enhancing pelvic floor muscle coordination.
2. Biofeedback: A behavior-based therapy with a feedback loop, enabling patients to visualize the impact of muscle actions and improve pelvic floor movements.
3. Rectal Balloon Training: Simulating resistance to the urge to defecate, aiding in LARS prevention.

   This will be carried out as in-person sessions weekly for the first month and biweekly for the next 2 months, totaling 8 sessions over 3 months. Additionally, home sessions will be conducted under phone guidance. Patients are required to fill out relevant questionnaires before and after completing the PFR program.

   The usual care group will receive standard post-surgical care.

   Baseline scores: Wexner's score, LARS score, EORTC CR 29 score taken before the start of the study.

   Follow-up: Participants will be followed for three months and Wexner's scores, LARS, EORTC CR 29 score will be taken.

   Quality Assurance

   Data Validation: Data entered into the registry will be validated against predefined rules for range and consistency.

   Source Data Verification: Data accuracy will be assessed by comparing registry data to external sources such as medical records.

   Data Dictionary: Detailed descriptions of each variable, including source, coding information, and normal ranges, will be maintained.

   Standard Operating Procedures (SOPs)

   Recruitment and Data Collection: SOPs will ensure consistent recruitment and data collection processes.

   Data Management and Analysis: Procedures for managing and analyzing data will be clearly defined.

   Adverse Event Reporting: SOPs will include protocols for reporting adverse events.

   Change Management: Procedures for handling changes in the study protocol will be in place.

   Sample Size Assessment:

   Previous Studies:

   Previous research has shown a reduction of Wexner's incontinence scores by 5 points (SD=8) with pelvic floor rehabilitation (PFR) treatment (6-9).

   Study Design:

   The study was designed with a significance level (alpha error or Type I error) set at 0.05 and a power of the test (beta error or Type II error) at 0.20. A total of 64 patients were initially calculated to be necessary to detect a statistically significant difference between treatment groups.

   Sample Size Calculation:

   Considering an anticipated drop-out rate of 20%, the total sample size required for the study was adjusted to 77 patients.

   Plan for Missing Data

   Procedures will be in place to address missing data, including how to handle variables reported as missing or inconsistent. We shall evaluate the extent of missing data for each variable and use appropriate methods for handling missing data such as imputation techniques or sensitivity analyses.

   Statistical Analysis Plan:

   Study Design

   The study involves a randomized controlled trial (RCT) where patients undergoing Sphincter sparing-rectal cancer surgery are randomized into two groups:

   Standard Group: Receives standard post-operative care. PFR Group: Receives pelvic floor physiotherapy in addition to standard care. Outcome Measures

   The following continuous variables will be measured before starting the intervention and after 3 months:

   Wexner's Scores: Assessing fecal incontinence severity. LARS Scores (Low Anterior Resection Syndrome): Assessing bowel dysfunction. EORTC CR 29 Scores (European Organisation for Research and Treatment of Cancer Colorectal Cancer Module): Assessing quality of life related to colorectal cancer.

   Statistical Hypotheses

   Within-Group Comparison:

   Null Hypothesis (H0): There is no significant difference in mean scores (Wexner's, LARS, EORTC CR 29) before and after intervention within each group (Standard and PFR).

   Between-Group Comparison:

   Null Hypothesis (H0): There is no significant difference in the change in mean scores (Wexner's, LARS, EORTC CR 29) from before to after intervention between the Standard and PFR groups.

   Statistical Methods

   Descriptive Statistics:

   Mean and standard deviation (SD) for continuous variables (Wexner's, LARS, EORTC CR 29 scores) at baseline and after 3 months in each group.

   Within-Group Analysis:

   Paired t-tests or Wilcoxon signed-rank tests (depending on normality) to compare mean scores before and after intervention within each group (Standard and PFR).

   Between-Group Analysis:

   Independent samples t-tests or Mann-Whitney U tests (depending on normality) to compare the change in mean scores (after - before) between the Standard and PFR groups.

   Adjustments:

   Adjustments for potential confounding factors such as age, gender, and baseline scores using analysis of covariance (ANCOVA) if necessary.

   Effect Size:

   Calculate effect sizes (e.g., Cohen's d for t-tests, r for Mann-Whitney U tests) to quantify the magnitude of differences observed.

   Statistical Significance:

   We shall set the significance level (alpha) at 0.05 to determine statistical significance.

   Software

   Utilize statistical software (SPSS) for data analysis. Reporting

   We shall present results with confidence intervals and p-values, providing clear interpretations of findings in relation to clinical significance and study objectives.

   This detailed description outlines the comprehensive approach taken to ensure the study's rigor and reliability, aiming to fill significant gaps in current knowledge about effective aftercare for rectal cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Age: Adults aged 18 years or older.
* Surgical Procedure: Have undergone Low Anterior Resection (LAR) for rectal cancer.
* Cognitive Ability: Capable of understanding and completing the questionnaires effectively

Exclusion Criteria:

* Medical History: History of proctitis, ulcerative colitis, or Crohn's disease.
* Surgical Extent: Extensive resection (beyond Total Mesorectal Excision - TME) for
* locally advanced (T4) tumors, patients undergoing APR.
* Surgical Complications: History of anastomotic leakage.
* Recent Physiotherapy: History of invasive physiotherapy within the past 6 months.
* Mental or Physical Inabilities: Inability to undergo Pelvic Floor Rehabilitation due to mental or physical limitations

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
WEXNER INCONTINENCE SCORE | Baseline score 6 weeks post-low anterior resection (LAR) or 6 weeks post-ileostomy closure. Post-intervention scores at 3 months post-start of pelvic floor physiotherapy for PFR group and 18 weeks post-LAR or post-ileostomy closure.
  The Wexner Incontinence Score assesses fecal incontinence severity using patient-reported symptoms. Scores range from 0 (no incontinence) to 20 (severe incontinence), with higher scores indicating worse outcomes. Patients evaluate bowel control, leakage frequency, and lifestyle impacts, providing crucial data for treatment evaluation and comparison in clinical trials.

SECONDARY OUTCOMES:
Low Anterior Resection Syndrome score (LARS) | Baseline score 6 weeks post-low anterior resection (LAR) or 6 weeks post-ileostomy closure. Post-intervention scores at 3 months post-start of pelvic floor physiotherapy for PFR group and 18weeks post-LAR or 18 weeks post-ileostomy closure.
  The LARS Score measures bowel dysfunction following low anterior resection surgery, with scores ranging from 0 to 42. Higher scores indicate more severe symptoms such as bowel movement frequency, urgency, and incontinence. This patient-reported outcome assesses the impact on daily life, guiding treatment strategies and evaluating post-surgical outcomes in clinical trials.
Quality of life measure QORTC CR 29 | Baseline score 6 weeks post-low anterior resection (LAR) or post-ileostomy closure. Post-intervention scores at 3 months post-start of pelvic floor physiotherapy for PFR group and 6 months post-LAR or 18 weeks post-ileostomy closure.
  The EORTC CR 29 assesses colorectal cancer-specific symptoms and treatment effects. Scores range from 0 to 100 per domain. Higher scores signify greater symptom burden or impact. Patients provide insights on bowel symptoms, urinary frequency, and emotional well-being, crucial for treatment assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Harshavardhana H P, MS DrNB (IP), Principal Investigator — GEM Coimbatore; RAJAPANDIAN S, DNB FRCS(Ed), Study Director — GEM Coimbatore; PALANIVELU C, MS Mch FRCS, Study Chair — GEM Coimbatore; HARISH KAKKILAYA, MS FACRSI, Study Director — GEM Coimbatore; SHANKAR B, MS DrNB FRCS, Study Director — GEM Coimbatore
Locations (1):
- GEM Hospital & Research Center, Coimbatore, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: Yes
We plan to share all individual participant data (IPD) that underlie the results reported in the publication. This includes de-identified data sets and relevant supporting documentation.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The IPD will be available 6 months after publication and will remain accessible for a period of 10 years.
Access Criteria: Access to the IPD will be granted to researchers who provide a methodologically sound proposal and are affiliated with academic institutions or research organizations. Requests will be reviewed by a data access committee based on scientific merit, feasibility, and ethical considerations. The review process will take approximately 4-6 weeks. Researchers can request access by submitting a proposal via our online application form. All researchers granted access will be required to sign a data use agreement to ensure responsible use of the data

REFERENCES:
- [Background] Lin KY, Granger CL, Denehy L, Frawley HC. Pelvic floor muscle training for bowel dysfunction following colorectal cancer surgery: A systematic review. Neurourol Urodyn. 2015 Nov;34(8):703-12. doi: 10.1002/nau.22654. Epub 2014 Aug 23. PMID 25156929
- [Background] Visser WS, Te Riele WW, Boerma D, van Ramshorst B, van Westreenen HL. Pelvic floor rehabilitation to improve functional outcome after a low anterior resection: a systematic review. Ann Coloproctol. 2014 Jun;30(3):109-14. doi: 10.3393/ac.2014.30.3.109. Epub 2014 Jun 23. PMID 24999460
- [Background] Maris A, Devreese AM, D'Hoore A, Penninckx F, Staes F. Treatment options to improve anorectal function following rectal resection: a systematic review. Colorectal Dis. 2013 Feb;15(2):e67-78. doi: 10.1111/codi.12036. PMID 23017030
- [Result] Camilleri-Brennan J, Ruta DA, Steele RJ. Patient generated index: new instrument for measuring quality of life in patients with rectal cancer. World J Surg. 2002 Nov;26(11):1354-9. doi: 10.1007/s00268-002-6360-2. Epub 2002 Sep 26. PMID 12297930
- [Result] Vironen JH, Kairaluoma M, Aalto AM, Kellokumpu IH. Impact of functional results on quality of life after rectal cancer surgery. Dis Colon Rectum. 2006 May;49(5):568-78. doi: 10.1007/s10350-006-0513-6. PMID 16583289
- [Result] Liu CH, Chen CH, Lee JC. Rehabilitation exercise on the quality of life in anal sphincter-preserving surgery. Hepatogastroenterology. 2011 Sep-Oct;58(110-111):1461-5. doi: 10.5754/hge11160. Epub 2011 Jul 15. PMID 21940307
- [Result] Allgayer H, Dietrich CF, Rohde W, Koch GF, Tuschhoff T. Prospective comparison of short- and long-term effects of pelvic floor exercise/biofeedback training in patients with fecal incontinence after surgery plus irradiation versus surgery alone for colorectal cancer: clinical, functional and endoscopic/endosonographic findings. Scand J Gastroenterol. 2005 Oct;40(10):1168-75. doi: 10.1080/00365520510023477. PMID 16165701
- [Result] Kim KH, Yu CS, Yoon YS, Yoon SN, Lim SB, Kim JC. Effectiveness of biofeedback therapy in the treatment of anterior resection syndrome after rectal cancer surgery. Dis Colon Rectum. 2011 Sep;54(9):1107-13. doi: 10.1097/DCR.0b013e318221a934. PMID 21825890
- [Result] Pucciani F, Ringressi MN, Redditi S, Masi A, Giani I. Rehabilitation of fecal incontinence after sphincter-saving surgery for rectal cancer: encouraging results. Dis Colon Rectum. 2008 Oct;51(10):1552-8. doi: 10.1007/s10350-008-9312-6. Epub 2008 May 2. PMID 18452041